CLINICAL TRIAL: NCT00285285
Title: A Randomized Trial to Assess the Efficacy of Point-of-Care Testing in Decreasing Length of Stay in a Pediatric Emergency Department
Brief Title: Point of Care Device Use in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Karen A. Santucci (Unknown); M. Douglas Baker (Unknown); i-Stat Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25448
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2006-01

CONDITIONS: Dehydration; Seizure; Gastroenteritis; Hyperglycemia
Keywords: Point-of-care Testing; Pediatric Emergency Department; Length of Stay; Efficiency
MeSH Terms: conditions — Dehydration; Seizures; Gastroenteritis; Hyperglycemia

INTERVENTIONS:
Device: Point of Care Device; i-Stat Analyzer

SUMMARY:
To compare the effect of "point-of-care" (POC) analysis of blood work with traditional laboratory methods on length of stay in a pediatric emergency department (PED).

DETAILED DESCRIPTION:
This study was a prospective, randomized controlled study of patients requiring blood work that a POC device was capable of performing. Length of time spent at various timepoints were prospectively recorded by a dedicated research assistant after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Clinically requiring bloodwork capable by the POC device

Exclusion Criteria:

* Requiring other bloodwork such as medication levels, WBC

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2004-01; Study Completion 2004-08

PRIMARY OUTCOMES:
Total Length of Stay

SECONDARY OUTCOMES:
Time length for results return, disposition decision, time in ED proper

CONTACTS AND LOCATIONS:
Overall Officials: M. Douglas Baker, MD, Study Director — Yale University